CLINICAL TRIAL: NCT07263295
Title: Evaluation of Diaphragmatic Function After Interscalene Brachial Plexus Block With Liposomal Bupivacaine: A Cohort Study
Brief Title: Evaluation of Diaphragmatic Function After Interscalene Block With Liposomal Bupivacaine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZJU_2025C116
Record Dates: First submitted 2025-09-27; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diaphragmatic Function; Metacarpal Fracture; Radius Fracture; Peripheral Nerve Neurolysis; Chronic Ulcer; Upper Extremity Ligament Injury
Keywords: Interscalene brachial plexus block; Liposomal Bupivacaine; Hemidiaphragmatic paralysis
MeSH Terms: conditions — Radius Fractures | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: 0.5% Hydrochloride Bupivacaine (10ml) + Liposomal Bupivacaine (10ml) for ISBPB (Experimental): ISBPB block group receiving combined administration of two drugs
  Interventions: Drug: 0.5% Hydrochloride Bupivacaine 10ml; Drug: Liposomal Bupivacaine 10mL
- 0.5% Hydrochloride Bupivacaine (20ml) for ISBPB (Active Comparator): ISBPB block control group receiving single administration of a single drug
  Interventions: Drug: 0.5% Hydrochloride Bupivacaine 20ml

INTERVENTIONS:
Drug: 0.5% Hydrochloride Bupivacaine 20ml — 0.5% Hydrochloride Bupivacaine 20ml for ISBPB
  Arms: 0.5% Hydrochloride Bupivacaine (20ml) for ISBPB
Drug: 0.5% Hydrochloride Bupivacaine 10ml — 0.5% Hydrochloride Bupivacaine 10ml for ISBPB
  Arms: Experimental Group: 0.5% Hydrochloride Bupivacaine (10ml) + Liposomal Bupivacaine (10ml) for ISBPB
Drug: Liposomal Bupivacaine 10mL — Liposomal Bupivacaine 10mL for ISBPB
  Arms: Experimental Group: 0.5% Hydrochloride Bupivacaine (10ml) + Liposomal Bupivacaine (10ml) for ISBPB

SUMMARY:
The study aims to evaluation the effects of Liposomal Bupivacaine on diaphragmatic function in patients undergoing upper limb surgery who receive Interscalene Brachial Plexus Block. A total of 120 eligible patients will be enrolled and divided into two groups: Group A will receive 20ml of 0.5% Hydrochloride Bupivacaine , while Group B will receive 10ml of 0.5% Hydrochloride Bupivacaine plus 10ml of Liposomal Bupivacaine. Assessments of diaphragmatic function, pulmonary function, and pain intensity will be performed before the block and at different time points after the block, with follow-up for adverse events. The study is scheduled to run from September 2025 to September 2026, with strict adherence to privacy protection and ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper limb surgery scheduled for interscalene brachial plexus block
* Aged ≥ 18 years
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Known allergy or intolerance to amide local anesthetics
* Nerve injury in the upper limb on the surgical side
* Coagulopathy
* Used opioid medications continuously for more than 3 weeks before surgery
* History of pulmonary disease and a pulse oxygen saturation (SpO₂) < 95% (measured after 5 minutes of rest at room temperature without oxygen supplementation, using a transcutaneous pulse oximeter)
* Refuse to participate or are deemed unsuitable for this trial by the researchers

Withdrawal Criteria:

* Patients voluntarily withdrew their informed consent
* Surgery was canceled or the anesthesia method was changed due to surgical factors before interscalene brachial plexus block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Identification the recovery time of diaphragmatic function after diaphragmatic paralysis caused by interscalene brachial plexus block | From the initiation of interscalene brachial plexus block to the recovery of diaphragmatic function (within approximately 72 hours)

SECONDARY OUTCOMES:
Identification the recovery time of pulmonary function after diaphragmatic paralysis | From the initiation of interscalene brachial plexus block to the recovery of pulmonary function (within approximately 72 hours)
Identification the Incidence of hemidiaphragmatic paralysis at different time points | From the initiation of interscalene brachial plexus block to the recovery of diaphragmatic function (within approximately 72 hours)
Identification the Proportion of pulmonary function recovery | Time Frame: From the initiation of interscalene brachial plexus block to the recovery of pulmonary function (within approximately 72 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, zhejiang 310000, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided